CLINICAL TRIAL: NCT03083613
Title: Phase II Trial of Raltitrexed and Paclitaxel as Second-line Chemotherapy for Patients With Unresectable or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: Raltitrexed and Paclitaxel for Gastric or Gastroesophageal Junction Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Aiping Zhou, Chief physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-G1-070
Record Dates: First submitted 2017-03-14; First posted 2017-03-20 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Adenocarcinoma
Keywords: Raltitrexed; Paclitaxel; chemotherapy; Gastric cancer; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms | interventions — raltitrexed; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Raltitrexed and Paclitaxel (Experimental): All patients receive the combination therapy of Raltitrexed and Paclitaxel for a maximum of 6 cycles
  Raltitrexed:3mg/m2,d1 Paclitaxel:80mg/m2,d1,d8,
  Eery 3 weeks
  Interventions: Drug: Raltitrexed; Drug: Paclitaxel

INTERVENTIONS:
Drug: Raltitrexed — Raltitrexed:3mg/m2,iv,d1, Every 3 weeks
  Other Names: RTX
Drug: Paclitaxel — Paclitaxel:80mg/m2,iv,d1,d8, Every 3 weeks

SUMMARY:
This is a single-arm clinical trial.The purpose of this study is to evaluate the efficacy and safety of Raltitrexed and Paclitaxel as second-line chemotherapy for patients with unresectable or metastatic gastric or gastroesophageal junction adenocarcinoma .The primary endpoint of this study is objective response rate.The secondary endpoint of this study is safety,progression-free survival and overall survival.

DETAILED DESCRIPTION:
Raltitrexed is an antifolate thymidylate synthase inhibitor that has shown efficacy and good safety profile in the treatment of colorectal cancer. To our knowledge, there has been no study published with the Raltitrexed and Paclitaxel regimen as second-line chemotherapy for patients with unresectable or metastatic gastric or gastroesophageal junction adenocarcinoma.The aim of our study was to evaluate the efficacy, safety and survival of this regimen in patients with unresectable or metastatic gastric or gastroesophageal junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed unresectable or metastatic gastric or gastroesophageal junction adenocarcinoma;
* Patients failed first-line chemotherapy containing fluoropyrimidines and platinums;
* ECOG (Eastern Cooperative Oncology Group)performance status 0-1;
* At least 1 measurable lesion should be present（RECIST1.1）
* Available Organ function: Neutrophils>2g/L, Hemoglobin>9g/L, Blood platelet >100g/L; Alanine aminotransferase(ALT） and Aspartate aminotransferase(AST)<1.5 ULN(upper limit of normal); Total bilirubin(TBIL)<1.0 ULN; Cr <1.0ULN
* Signed informed consent.
* Life expectancy ≥3 months;

Exclusion Criteria:

* Previous treatment with Raltitrexed or Paclitaxel;
* Known history of allergic reaction to Raltitrexed or Paclitaxel;
* Known brain metastases;
* Pregnant or breast feeding women;
* Severe diarrhea,intestinal obstruction;
* other co-existing malignancies or malignancies diagnosed within the last 5 years(except cured cutaneum carcinoma or carcinoma in situs of cervix);
* Previous myocardial infarction, unstable angina, stroke ,or uncontrollable Arrhythmia;
* Kown HIV infecton.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-05; Primary Completion 2017-09-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | 18-26 months

SECONDARY OUTCOMES:
Overall Survival | 18-26 months
  From date of randomization until date of death
Progression-free survival | 18-26 months
  From date of randomization until date of first documented PD, date of death

CONTACTS AND LOCATIONS:
Overall Officials: Ai Ping Zhou, Doctor of medcine, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No